CLINICAL TRIAL: NCT05153564
Title: Investigation of the Effect of Subcutaneously Co-administered Semaglutide and NNC0480-0389 on Pharmacokinetics of an Oral Combination Contraceptive (Ethinylestradiol and Levonorgestrel) in Healthy Postmenopausal Females
Brief Title: A Research Study Looking Into the Effect of Semaglutide and NNC0480 0389 on Blood Levels of a Birth Control Pill in Woman After Menopause
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9389-4681; 2021-003060-27 (EudraCT Number); U1111-1266-3910 (Other: WHO)
Record Dates: First submitted 2021-12-08; First posted 2021-12-10 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One-sequence cross-over arm (Experimental)
  Interventions: Drug: Semaglutide 1.34 mg/mL; Drug: Semaglutide 3.0 mg/mL; Drug: NNC0480-0389 10 mg/mL; Drug: NNC0480-0389 30 mg/mL; Drug: Microgynon®

INTERVENTIONS:
Drug: Semaglutide 1.34 mg/mL — Semaglutide will be administered at a dose of 0.25, 0.50 or 1.0 mg as indicated on scale drum once weekly by subcutaneous (s.c.) (under the skin) injections in the abdomen for 14 weeks.
Drug: Semaglutide 3.0 mg/mL — Semaglutide will be administered at a dose of 2.0 mg corresponding to the increment of 67 (pen injector units) as indicated on scale drum. once weekly by subcutaneous (s.c.) (under the skin) injections in the abdomen for 14 weeks.
Drug: NNC0480-0389 10 mg/mL — NNC0480-0389 will be administered at a dose of 0.23, 0.45 or 0.90 mL once weekly by s.c. (under the skin) injections for 14 weeks.
Drug: NNC0480-0389 30 mg/mL — NNC0480-0389 will be administered at a dose of 0.60 mL once weekly by s.c. (under the skin) injections for 14 weeks.
Drug: Microgynon® — Microgyn® will be given as once daily oral dosing in two periods, each of 8 days' duration. One tablet contains levonorgestrel 0.15 mg and ethinylestradiol 0.03 mg.

SUMMARY:
Novo Nordisk is developing a combination therapy with the investigational drug NNC0480-0389 and an already approved medicine called "semaglutide" for the treatment of type-2 diabetes (T2D). It is expected that the combination will further improve the blood sugar control compared to semaglutide therapy alone. The study will investigate the influence of the combination of semaglutide and NNC0480-0389 on the blood levels of a birth control pill (a combined oral contraceptive consisting of ethinylestradiol and levonorgestrel) and paracetamol. Participants will get semaglutide and NNC0480-0389 as injection under the skin of their belly using a pen-injector. The injections will be given once weekly for 14 weeks. Additionally, participants will at two occasions get paracetamol as soluble tablet in connection with a standardised breakfast meal. Further, participants will get the birth control pill in form of tablets in two periods of 8 days each. Participants will get the combination of semaglutide and NNC0480-0389 as well as paracetamol and the combined contraceptive in any case. The study participation will last up to about 24 weeks. Participants will have 25 visits at the study centre. For 4 of the visits participants will stay at the study centre; the remaining visits will be outpatient. Only healthy postmenopausal women can take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, aged greater than or equal to 45 years at the time of signing informed consent
* Body mass index between 20.0 and 29.9 kilogram per meter square (kg/m^2) (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* HbA1c greater than or equal to 6.5 % (48 millimoles per mole (mmol/mol)) at screening
* Use of prescription medicinal products or non-prescription drugs including any herbal medicine known to interfere with the metabolic cytochrome P450 enzyme (CYP) pathways, such as hypericum (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae, within 14 days before screening. Exceptions are routine vitamins, occasional use of paracetamol, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation
* Use of hormone replacement therapy within 4 weeks before first dose of trial product or intention to initiate treatment with hormone replacement therapy during the study
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Area under the ethinylestradiol plasma concentration time curve during a dosing interval (0 to 24 hours) at steady state (AUC0-24h,EE,SS) | From pre-dose to 24 hours after last dosing of oral contraceptive on day 8 and day 100
  Measured in h*pg/mL
Area under the levonorgestrel plasma concentration time curve during a dosing interval (0 to 24 hours) at steady state (AUC0-24h,LN,SS) | From pre-dose to 24 hours after last dosing of oral contraceptive on day 8 and day 100
  Measured in h*pg/mL

SECONDARY OUTCOMES:
Maximum concentration of ethinylestradiol at steady state (Cmax,EE,SS) | Within pre-dose to 24 hours after last dosing of oral contraceptive on day 8 and day 100
  Measured in pg/mL
Maximum concentration of levonorgestrel at steady state (Cmax,LN,SS) | Within pre-dose to 24 hours after last dosing of oral contraceptive on day 8 and day 100
  Measured in pg/mL
Area under the paracetamol concentration-time curve for 0-60 minutes following a standardised meal (AUC0-60min,para) | From pre-dose to 60 minutes after dosing of paracetamol on day 1 and day 93
  Measured in h*μg/mL
Area under the paracetamol concentration-time curve for 0-300 minutes following a standardised meal (AUC0-300min,para) | From pre-dose to 300 minutes after dosing of paracetamol on day 1 and day 93
  Measured in h*μg/mL
Maximum observed paracetamol concentration following a standardised meal (Cmax,para) | Within pre-dose to 300 minutes after dosing of paracetamol on day 1 and day 93
  Measured in μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com